CLINICAL TRIAL: NCT00002549
Title: RANDOMIZED PHASE III STUDY OF INDUCTION (ICE VS MICE VS DCE) AND INTENSIVE CONSOLIDATION (IDIA VS NOVIA VS DIA) FOLLOWED BY BONE MARROW TRANSPLANTATION IN ACUTE MYELOGENOUS LEUKEMIA: AML 10 PROTOCOL
Brief Title: Combination Chemotherapy Followed by Bone Marrow or Peripheral Stem Cell Transplantation in Treating Patients With Acute Myelogenous Leukemia
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000063311; EORTC-06931
Record Dates: First submitted 1999-11-01; First posted 2004-07-19 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Leukemia
Keywords: untreated adult acute myeloid leukemia; adult acute erythroid leukemia (M6); adult acute myeloblastic leukemia without maturation (M1); adult acute myeloblastic leukemia with maturation (M2); adult acute myelomonocytic leukemia (M4); adult acute monoblastic leukemia (M5a); adult acute megakaryoblastic leukemia (M7); secondary acute myeloid leukemia; adult acute monocytic leukemia (M5b)
MeSH Terms: conditions — Leukemia; Leukemia, Erythroblastic, Acute; Leukemia, Myeloid, Acute; Leukemia, Myelomonocytic, Acute; Leukemia, Monocytic, Acute; Leukemia, Megakaryoblastic, Acute | interventions — Filgrastim; Busulfan; Cyclophosphamide; Cytarabine; Daunorubicin; Etoposide; Idarubicin; Mesna; Mitoxantrone; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Biological: filgrastim
Drug: busulfan
Drug: cyclophosphamide
Drug: cytarabine
Drug: daunorubicin hydrochloride
Drug: etoposide
Drug: idarubicin
Drug: mesna
Drug: mitoxantrone hydrochloride
Procedure: allogeneic bone marrow transplantation
Procedure: autologous bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Combining chemotherapy with peripheral stem cell or bone marrow transplantation may allow the doctor to give higher doses of chemotherapy drugs and kill more cancer cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of combination chemotherapy followed by bone marrow or peripheral stem cell transplantation in treating patients with acute myelogenous leukemia.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the complete remission (CR) rate following 1 or 2 courses of ICE (idarubicin/cytarabine/etoposide) vs. MICE (mitoxantrone/cytarabine/etoposide) vs. DCE (daunorubicin/cytarabine/etoposide) in patients with newly diagnosed acute myeloid leukemia. II. Compare disease-free survival and overall survival achieved with each anthracycline on the above induction regimens and with intermediate-dose cytarabine (IDIA vs. NOVIA vs. DIA) as consolidation therapy. III. Compare disease-free survival, relapse rate, death in first CR, and overall survival in patients who receive peripheral blood stem cells (PBSC) vs. autologous bone marrow transplant (AuBMT) vs. allogeneic bone marrow transplant (AlBMT) as rescue from myeloablative therapy following remission consolidation. IV. Assess the time to recovery of normal or acceptable polymorphonuclear leukocyte and platelet counts following each treatment step. V. Determine the incidence and type of grade 4 toxicity and treatment-related mortality. VI. Evaluate the quality of life during each step of treatment using self-administered questionnaires. VII. Compare stem cell mobilization after IDIA vs. NOVIA vs. DIA, each using granulocyte colony-stimulating factor as the mobilizing growth factor. VIII. Assess the rate of completion of stem cell transplantation using PBSC vs. AlBMT vs. AuBMT as the last step of therapy. IX. Compare the costs of treatment (e.g., antibiotics and transfusion requirements) and hospitalization duration between the AuBMT vs. PBSC.

OUTLINE: Randomized study. All patients are randomized to Arms I, II, and III for Induction/Consolidation. Patients in CR following Consolidation who have an HLA-identical sibling, are less than 45 or 55 years of age (depending on center policy), and have adequate organ function are nonrandomly assigned to AlBMT on Regimen A; those in CR who are without an available sibling donor and who have adequate organ function proceed to Regimen B, then are randomized to Arms IV and V. The following acronyms are used: AlBMT Allogeneic Bone Marrow Transplant ARA-C Cytarabine, NSC-63878 AuBMT Autologous Bone Marrow Transplant BU Busulfan, NSC-750 CTX Cyclophosphamide, NSC-26271 DCE DNR/ARA-C/VP-16 DHAD Mitoxantrone, NSC-301739 DIA DNR/ID ARA-C DNR Daunorubicin, NSC-82151 G-CSF Granulocyte Colony-Stimulating Factor (Rhone-Poulenc-Rorer) ICE IDA/ARA-C/VP-16 IDA Idarubicin, NSC-256439 ID Intermediate Dose IDIA IDA/ID ARA-C Mesna Mercaptoethane sulfonate, NSC-113891 MICE DHAD/ARA-C/VP-16 NOVIA DHAD/ID ARA-C PBSC Peripheral Blood Stem Cells TBI Total-Body Irradiation VP-16 Etoposide, NSC-141540 INDUCTION/CONSOLIDATION: Arm I: 3-Drug Combination Chemotherapy followed by 2-Drug Combination Chemotherapy. ICE; followed by IDIA. Arm II: 3-Drug Combination Chemotherapy followed by 2-Drug Combination Chemotherapy. MICE; followed by NOVIA. Arm III: 3-Drug Combination Chemotherapy followed by 2-Drug Combination Chemotherapy. DCE; followed by DIA. POSTCONSOLIDATION THERAPY: Regimen A: Single-Agent Chemoablation plus Radioablation or 2-Drug Chemoablation followed by Hematopoietic Rescue. CTX; plus TBI (equipment unspecified); or CTX/BU; followed by AlBMT. Entry on EORTC study comparing CI IDA with standard CTX/TBI or CTX/BU encouraged. Regimen B: Stem cell Mobilization and Harvest. G-CSF or CTX/G-CSF. Arm IV: Single-Agent Chemoablation plus Radioablation or 2-Drug Chemoablation followed by Hematopoietic Rescue. CTX/TBI or CTX/BU; followed by PBSC. Arm V: Single-Agent Chemoablation plus Radioablation or 2-Drug Chemoablation followed by Hematopoietic Rescue. CTX/TBI or CTX/BU; followed by AuBMT.

PROJECTED ACCRUAL: 1,520 patients will be randomized for Induction/Consolidation over about 5 years; if excessive deaths are found at interim analyses, the inferior arm will close. It is expected that 744 patients will be randomized for Postconsolidation therapy, with 345 patients followed until relapse/death.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Newly diagnosed acute myeloid leukemia (AML) of any FAB histology (M1-M7) except M3 At least 30% blast cells in bone marrow smears Secondary leukemias eligible, as follows: Following cured malignancies, including Hodgkin's disease Following exposure to alkylating agents or radiotherapy for other reasons The following leukemias are excluded: Blast crisis of chronic myeloid leukemia Leukemia secondary to other myeloproliferative disease Leukemia secondary to myelodysplastic syndrome of more than 6 months' duration No other progressive malignant disease

PATIENT CHARACTERISTICS: Age: 15 to 60 Performance status: Not specified Hematopoietic: Not applicable Hepatic: Bilirubin no greater than 1.5 x ULN Renal: Creatinine no greater than 1.5 x ULN Cardiovascular: No severe heart failure requiring diuretics or with an LVEF less than 50% Other: No severe concomitant neurologic disease No severe concomitant psychologic disease

PRIOR CONCURRENT THERAPY: No prior therapy for AML (chemotherapy, radiotherapy, or more than 7 days of corticosteroids)

Ages: 15 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1520 (Estimated)
Dates: Start 1993-11

CONTACTS AND LOCATIONS:
Overall Officials: Robert A. Zittoun, MD, Study Chair — Hotel Dieu de Paris
Locations (75):
- Universitaetsklinik, Innsbruck, Austria
- Belgium (6):
  - Algemeen Ziekenhuis Middelheim, Antwerp
  - A.Z. St. Jan, Bruges
  - Hopital Universitaire Erasme, Brussels
  - Institut Jules Bordet, Brussels (Bruxelles)
  - Universitair Ziekenhuis Antwerpen, Edegem
  - CHU Sart-Tilman, Liège
- Croatia (2):
  - University Hospital Rebro, Zagreb
  - Medical School/University of Zagreb, Zagreb (Agram)
- Czechia (2):
  - University Hospital - Olomouc, Olomouc
  - Institute of Hematology and Blood Transfusion, Prague
- France (7):
  - Hopital Edouard Herriot, Lyon
  - Centre Antoine Lacassagne, Nice
  - Hotel Dieu de Paris, Paris
  - Hopital Cochin, Paris
  - Hopital Necker, Paris
  - Centre Medico-Chirurgical Foch, Suresnes
  - Institut Gustave Roussy, Villejuif
- Germany (2):
  - Staedtische Kliniken Duisburg, Duisburg
  - Klinikum Grosshadern, Munich (Muenchen)
- County Hospital, Kecskemét, Hungary
- Italy (45):
  - Ospedale Civile Alessandria, Alessandria
  - Ospedale Torrette University Ancona, Ancona
  - Ospedale Civile Avellino, Avellino
  - Universita Degli Studi di Bari Policlinico, Bari
  - Ospedale Regionale A. Di Summa, Brindisi
  - Ospedale Oncologico A. Businco, Cagliari
  - Ospedale Ferrarotto, Catania
  - Ospedale Regionale A. Pugliese, Catanzaro
  - Centro Trapianti di Midollo Osseo, Cremona
  - Ospedale Santa Croce, Cuneo
  - Universita Degli Studi di Firenze - Policlin. di Careggi, Firenze (Florence)
  - Ospedali Riuniti Foggia, Foggia
  - Ospedale S. Antonio Abate, Gallarate Varese
  - Ospedale San Martino/Cliniche Universitarie Convenzionale, Genoa (Genova)
  - Ospedale Gen. Provinciale Santa Maria Goretti, Latina
  - Ospedale Maggiore Lodi, Lodi
  - Instituto Scientifico H.S. Raffaele, Milano (Milan)
  - Ospedale Maggiore Ca Granda, Milano (Milan)
  - Universita di Modena, Modena
  - Azienda Ospedaliera "A. Cardarelli", Naples (Napoli)
  - Federico II University Medical School, Naples (Napoli)
  - Ospedale S. Gennora USL 42, Naples (Napoli)
  - Ospedale Nuovo Pellegrini, Naples (Napoli)
  - Ospedale Maggiore, Novara
  - Ospedale San Francesco, Nuoro
  - Azienda Ospedale S. Luigi - Universita Di Torino, Orbassano, (Torino)
  - Policlinico - Cattedra di Ematologia, Palermo
  - Policlinico P. Giaccone - Universita Di Palermo, Palermo
  - Ospedale Cervello, Palermo
  - Azienda Ospedaliera Di Parma, Parma
  - University and I.R.C.C.S. Policlinico San Matteo, Pavia
  - Policlinico Monteluce, Perugia
  - Ospedale San Salvatore, Pesaro
  - Ospedale Civile Pescara, Pescara
  - Ospedale San Carlo, Potenza
  - Ospedali Riuniti, Reggio Calabria
  - Arcispedale S. Maria Nuova, Reggio Emilia
  - Ospedale San Eugenio, Rome
  - Azienda Policlinico Umberto Primo, Rome
  - Policlinico A. Gemelli - Universita Cattolica del Sacro Cuore, Rome
  - Ospedale Casa Sollievo della Sofferenza, San Giovanni Rotondo
  - Istituto di Ematologia Universita - University di Sassari, Sassari
  - Azienda Ospedaliera Ospedale E. Mortelli, Sondalo (so)
  - Ospedal SS Annunziata, Taranto
  - Ospedale Molinette, Turin (Torino)
- Netherlands (6):
  - Groot Ziekengasthuis 's-Hertogenbosch, 's-Hertogenbosch
  - Onze Lieve Vrouwe Gasthuis, Amsterdam
  - Medisch Spectrum Twente, Enschede
  - Leiden University Medical Center, Leiden
  - University Medical Center Nijmegen, Nijmegen
  - Sint Joseph Ziekenhuis, Veldhoven
- Portugal (2):
  - Hospitais da Universidade de Coimbra (HUC), Coimbra
  - Hospital Escolar San Joao, Porto
- Ibn-i Sina Hospital, Ankara Univeristy, Ankara, Turkey (Türkiye)

REFERENCES:
- [Background] Maurillo L, Buccisano F, Spagnoli A, et al.: In acute myeloid leukemia, the use in induction of standard dose arac is associated with a better quality of response as compared to an induction regimen containing high dose arac. [Abstract] Blood 114 (22): A-1584, 2009.
- [Background] Oosterveld, M, Suciu S, Muus P, et al.: A new prognostic disease specific model to predict survival after intensive antileukemic treatment for young patients with poor-risk MDS and AML: results of the CRIANT and AML-10 studies conducted by the EORTC/GIMEMA/SAKK/HOVON/EBMT groups. [Abstract] Blood 104 (11): A-2020, 2004.
- [Result] Mandelli F, Vignetti M, Suciu S, Stasi R, Petti MC, Meloni G, Muus P, Marmont F, Marie JP, Labar B, Thomas X, Di Raimondo F, Willemze R, Liso V, Ferrara F, Baila L, Fazi P, Zittoun R, Amadori S, de Witte T. Daunorubicin versus mitoxantrone versus idarubicin as induction and consolidation chemotherapy for adults with acute myeloid leukemia: the EORTC and GIMEMA Groups Study AML-10. J Clin Oncol. 2009 Nov 10;27(32):5397-403. doi: 10.1200/JCO.2008.20.6490. Epub 2009 Oct 13. PMID 19826132
- [Derived] Baron F, Stevens-Kroef M, Kicinski M, Meloni G, Muus P, Marie JP, Halkes CJM, Thomas X, Vrhovac R, Albano F, Lefrere F Sr, Sica S, Mancini M, Venditti A, Hagemeijer A, Jansen JH, Amadori S, de Witte T, Willemze R, Suciu S. Impact of induction regimen and allogeneic hematopoietic cell transplantation on outcome in younger adults with acute myeloid leukemia with a monosomal karyotype. Haematologica. 2019 Jun;104(6):1168-1175. doi: 10.3324/haematol.2018.204826. Epub 2018 Dec 6. PMID 30523055
- [Derived] Baron F, Stevens-Kroef M, Kicinski M, Meloni G, Muus P, Marie JP, Halkes CJM, Thomas X, Vrhovac R, Specchia G, Lefrere F Sr, Sica S, Mancini M, Venditti A, Hagemeijer A, Becker H, Jansen JH, Amadori S, de Witte T, Willemze R, Suciu S. Cytogenetic clonal heterogeneity is not an independent prognosis factor in 15-60-year-old AML patients: results on 1291 patients included in the EORTC/GIMEMA AML-10 and AML-12 trials. Ann Hematol. 2018 Oct;97(10):1785-1795. doi: 10.1007/s00277-018-3396-4. Epub 2018 Jun 20. PMID 29926156